CLINICAL TRIAL: NCT02665364
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Neutralization of the Interferon Gene Signature and the Clinical Efficacy of IFNα-Kinoid in Adult Subjects With Systemic Lupus Erythematosus
Brief Title: Phase IIb Study of IFN-K in Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reorganization proceedings of the sponsor
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFN-K-002
Record Dates: First submitted 2015-11-17; First posted 2016-01-27 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — montanide ISA 51

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IFNα-Kinoid (Experimental): IFNα-Kinoid (IFN-K) adjuvanted with ISA 51 VG via intramuscular injection. 1 administration of 240 μg at W0, W1, W4 and 1 administration of 120 μg at month 3 (W12) and month 6 (W24) in addition to standard of care treatment.
  Interventions: Biological: IFNα-Kinoid; Other: ISA 51 VG
- Placebo (Placebo Comparator): Placebo normal saline (0.9% Sodium Chloride) adjuvanted with ISA 51 VG via intramuscular injection. 1 administration of 240 μg at week (W)0, W1, W4 and 1 administration of 120 μg at month 3 (W12) and month 6 (W24) in addition to standard of care treatment.
  Interventions: Other: Placebo; Other: ISA 51 VG

INTERVENTIONS:
Biological: IFNα-Kinoid
  Arms: IFNα-Kinoid
Other: Placebo
  Arms: Placebo
Other: ISA 51 VG

SUMMARY:
The safety and immunogenicity of the IFNα-Kinoid (IFN-K) have been evaluated in a phase I clinical study conducted in subjects with Systemic Lupus Erythematosus (SLE). Preliminary results showed acceptable safety profile and patients developped antibodies response.

The principal aim of the present study is to confirm the neutralization of the interferon gene signature and the clinical efficacy of IFN-K in subjects with SLE. In addition, the immune responses and the safety elicited by IFN-K will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has had a diagnosis of SLE according to current American College of Rheumatology (ACR) criteria (4 of 11 ACR criteria)
* Has SLEDAI-2K ≥ 6
* Has at least 1 BILAG A and/or at least 2 BILAG B
* Has a positive IFN gene signature by reverse transcription quantitative polymerase chain reaction (RT-qPCR)
* Has anti-nuclear antibodies (ANA) ≥ 1:160 and/or anti-dsDNA antibodies ≥ 7.0 IU/mL
* Currently receiving at least one treatment for SLE

Exclusion Criteria:

* Has active, severe lupus nephritis as defined either by the immediate need for cyclophosphamide treatment or by renal BILAG A
* Has active, severe, neuropsychiatric SLE, defined as neuropsychiatric BILAG A
* Has been treated with corticosteroids (CS) at a dose of >20 mg of prednisone equivalent/day for > 7 consecutive days
* Is currently receiving or has received pulse dose CS (≥ 250 mg prednisone equivalent/day)
* Has received potent immunosuppressive drugs
* Has received abatacept, sifalimumab, rontalizumab, anifrolumab, belimumab, tumor necrosis factor (TNF) antagonists or another registered or investigational biological therapy
* Has received anti-B-cell therapy (e.g., rituximab, epratuzumab)
* Has frequent recurrences of oral or genital herpes simplex lesions
* Is at high risk of significant infection and/or has any current signs or symptoms of infection at entry or has received intravenous antibiotics
* Has received any live vaccine
* Has used any investigational or non-registered product or any investigational or non-registered vaccine
* Is high-risk human papilloma virus (HPV) positive by rRT-qPCR on a cervical swab
* Has cytological abnormalities ≥ high grade squamous intraepithelial lesions (HSIL) on a cervical swab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Houssiau, MD, PhD, Study Chair — Head of Rhumatology, UCL, Brussels, Belgium
Locations (71):
- United States (11):
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Charlotte, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Austin, Texas
- Research Site, Buenos Aires, Argentina
- Research Site, Brussels, Belgium
- Research Site, Santiago, Chile
- Colombia (5):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Zipaquirá
- Research Site, Zagreb, Croatia
- France (6):
  - Research Site, Pessac, Bordeaux
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research site, Strasbourg
- Research Site, Tbilisi, Georgia
- Germany (5):
  - Research site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, Munich
- Italy (6):
  - Research Site, Rome, Roma
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Verona
- Mexico (4):
  - Research Site, Cuernavaca
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, México
- Research Site, Chisinau, Moldova
- Research Site, Lima, Peru
- Philippines (4):
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Manila
  - Research Site, Quezon
- Poland (7):
  - Research Site, Bytom
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Sosnowiec
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (8):
  - Research Site, Chelyabinsk
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Yekaterinburg
- Research Site, Seoul, South Korea
- Research Site, Lausanne, Switzerland
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Research Site, Bangkok, Thailand
- Tunisia (3):
  - Research Site, Sfax
  - Research Site, Sousse
  - Research Site, Tunis

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Houssiau FA, Thanou A, Mazur M, Ramiterre E, Gomez Mora DA, Misterska-Skora M, Perich-Campos RA, Smakotina SA, Cerpa Cruz S, Louzir B, Croughs T, Tee ML. IFN-alpha kinoid in systemic lupus erythematosus: results from a phase IIb, randomised, placebo-controlled study. Ann Rheum Dis. 2020 Mar;79(3):347-355. doi: 10.1136/annrheumdis-2019-216379. Epub 2019 Dec 23. PMID 31871140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants enrolled is the number of participants who signed informed condent form.
  One subject was randomized in IFN-K group and did not receive IFN-K. A total of 185 subjects were randomized and 184 subjects were treated : 91 subjects received IFN-K and 93 subjects received placebo.
Groups:
- IFN-K: Subjects received IFN-K adjuvanted with ISA 51 VG via intramuscular injection. 1 administration of 240 μg at W0, W1, W4 and 1 administration of 120 μg at month 3 (W12) and month 6 (W24) in addition to standard of care treatment.
- Placebo: Subjects received placebo normal saline (0.9% Sodium Chloride) adjuvanted with ISA 51 VG via intramuscular injection. 1 administration of 240 μg at week (W)0, W1, W4 and 1 administration of 120 μg at month 3 (W12) and month 6 (W24) in addition to standard of care treatment.
Period: Overall Study
Arm/Group | IFN-K | Placebo
Started | 91 | 93
Completed | 85 | 84
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Population: A total of 185 subjects were randomized. One subject was randomized in IFN-K group and did not receive IFN-K. 184 subjects were treated; 91 subjects received IFN-K and 93 subjects received placebo.
Groups:
- IFN-Kinoid: IFN-K adjuvanted with ISA 51 VG
- Placebo: Placebo adjuvanted with ISA 51 VG
- Total: Total of all reporting groups
Arm/Group | IFN-Kinoid | Placebo | Total
Number analyzed (Participants) | 91 | 93 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 93 | 184
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 88 | 172
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Eyhnic origin: Black | 1 | 1 | 2
  Eyhnic origin: Asian | 16 | 10 | 26
  Eyhnic origin: Caucasian/Hispanic | 68 | 72 | 140
  Eyhnic origin: Other | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  Colombia | 9 | 9 | 18
  United States | 2 | 4 | 6
  Philippines | 10 | 9 | 19
  Moldova | 6 | 14 | 20
  Thailand | 3 | 0 | 3
  Russia | 9 | 13 | 22
  South Korea | 1 | 0 | 1
  Belgium | 1 | 0 | 1
  Taiwan | 1 | 1 | 2
  Poland | 13 | 5 | 18
  Italy | 3 | 3 | 6
  Mexico | 10 | 9 | 19
  Georgia | 2 | 3 | 5
  France | 1 | 0 | 1
  Chile | 2 | 4 | 6
  Peru | 10 | 11 | 21
  Germany | 2 | 2 | 4
  Croatia | 1 | 1 | 2
  Argentina | 0 | 1 | 1
  Tunisia | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in IFN Gene Signature at W36
Description: The biological endpoint aimed at evaluating the neutralization of the IFN gene signature following treatment with IFN-K compared to placebo, as measured by the % change from baseline of the expression of IFN-induced genes.
Time Frame: Baseline and Last Available Value (LVA) between week 24 and week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 87 had a Last available value (LAV) between Week 24 and Week 36 analyzed. 93 subjects received placebo, among them, 84 had LAV between Week 24 and Week 36 analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- IFN-K: IFN-K adjuvanted with ISA 51 VG
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 87 | 84
percent change | -31.04 (38.96) | -0.44 (27.34)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; The percent of change from baseline to last available value between W24 and W36 of treatment in the expression of IFN-induced genes was analyzed using an analysis of covariance (ANCOVA) model; Test type: Superiority; p < 0.0001, ANCOVA; arithmetic mean = -30.2802, 95% CI 2-sided [-40.6653 to -19.8951], Standard Error of Mean 5.2588

2. Primary Outcome: Number of Participants Who Achieved a British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) With Superimposed CS Tapering at Week 36
Description: British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) responder was defined as a subject who had the following criteria at week 36:
  * All BILAG A scores at baseline improve to B/C/D and all BILAG B scores improve to C/D at W36, and
  * No BILAG worsening in other body systems: no new BILAG A or ≥ 2 new BILAG B scores at W36, and
  * No worsening in SLEDAI-2K total score at W36 compared with baseline, and
  * No deterioration in Physician Global Assessment (PGA) (< 10% worsening) on Visual Analog Scale (VAS) 100 mm at W36 compared with baseline, and
  * No addition or increased dose level of anti-malarial drugs or immunosuppressive drugs or CS* between W24 and W36 (*≤5 mg prednisolone or equivalent /day at W24 and no increase until W36).
Time Frame: At Week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 85 completed Week 36 visit. 93 subjects received placebo, among them, 84 completed Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 85 | 84
Participants | 35 | 29
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Descriptive statistics for the response to treatment according to BICLA at week 36 were presented by treatment group. The response to treatment according to BICLA was analyzed using a logistic regression with the response rate as dependent variable and treatment as independent variable, while adjusting for the minimization factors used for randomization; Test type: Superiority; p = 0.34, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.716 to 2.657]

3. Secondary Outcome: Number of Participants Who Achieved a Systematic Lupus Erythematosus (SLE) Responder Index (SRI)-4 at Week 36
Description: SLE Responder Index (SRI); SRI-4 responder was defined as a subject who had the following criteria at week 36:
  * reduction ≥4 points in SELENA-SLEDAI at week 36 compared with baseline, and
  * no new BILAG A at week 36, and
  * no more than 1 new BILAG B at week 36, and
  * no deterioration in PGA (<10% worsening) on 100-mm VAS compared with baseline
Time Frame: W36 (9 months)
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 84 completed Week 36 visit. 93 subjects received placebo, among them, 83 completed Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 84 | 83
Participants | 57 | 54
Statistical Analysis 1: Comparison: IFN-K vs Placebo; The SRI-4 response was analyzed using a logistic regression using the response rate as dependent variable and treatment as independent variable, while adjusting for the minimization factors used for randomization; Test type: Superiority; p = 0.6243, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.602 to 2.329]

4. Secondary Outcome: Number of Participants Who Achieved a Lupus Low Disease Activity State (LLDAS) at Week 36
Description: Lupus low disease activity state (LLDAS) was conceptually defined as 'a state which, if sustained, is associated with a low likelihood of adverse outcome, considering disease activity and medication safety'. Subsequently defined using consensus methodology, LLDAS is attained if all the following items are met:
  * SLEDAI-2K ≤4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity
  * No new features of lupus disease activity compared with the previous assessment
  * SELENA-SLEDAI physician global assessment (PGA, scale 0-3) ≤1
  * Current prednisolone (or equivalent) dose ≤7.5 mg daily
  * Well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents, excluding investigational drugs
Time Frame: At Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 85 | 84
Participants | 45 | 25
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0022, Pearson's Chi-squared

5. Secondary Outcome: BILAG Global Score Change From Baseline to Last Available Value (LVA) Between Week 24 and Week 36
Description: British Isles Lupus Assessment Group (BILAG)-2004 index, it categorizes disease activity into 5 different levels from A to E, with Grade A representing very active disease and Grade E indicating no current or previous disease activity. Scoring was based on a total of 101 items, grouped into 9 organ/systems and the summation of the numerical values for the nine-system scores was given by the following formula: Numerical global score = A*12 + B*8 + C*1, where A, B and C represent the number of Grades A, B and C respectively at each assessment. Grades D and E are considered as 0 (Chee-Seng Yee et al, 2010). The minimum score is 0 with no predefined maximum. The higher scores mean a worse outcome.
  The BILAG global score change from baseline to Last Available Value (LVA) week 24 and week 36 were presented analyzed.
Time Frame: Last Available Value (LVA) between week 24 and week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 87 | 84
scores on a scale | -11.43 (8.57) | -10.76 (7.84)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Baseline to last available value between W24 and W36; Test type: Superiority; p = 0.7946, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: SELENA-SLEDAI - Change From Baseline to Week 36
Description: Safety of Estrogens in Systemic Lupus Erythematosus National Assessment (SELENA)-SLEDAI, is a slightly modified version of the SLEDAI. This is a weighted index in which signs and symptoms, laboratory tests, and Physician's Global Assessment (PGA) for each of nine organ systems are given a weighted score and summed up if present at the time of the visit or in the preceding 10 days. The maximum theoretical score for the SELENA SLEDAI is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease.
Time Frame: Baseline and Week 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SELENA SLEDAI Score
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 84 | 83
SELENA SLEDAI Score | -5.48 (4.30) | -5.54 (4.44)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.9224, student - pooled

7. Secondary Outcome: SLICC/ACR-DI Change From Baseline at Week 36
Description: Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index for systemic lupus erythematosus (SLICC/ACR-DI) captures permanent changes which have occurred in patients with SLE, regardless of causality. The questionnaire contains 41 items covering 12 different organ systems. The score of items ranges from 1 to 3 and the total score from 0 to 47. By definition score 0 corresponds to diagnostics and damage over time can only be stable or increase, theoretically to a maximum of 47 points.
Time Frame: Baseline and Week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 82 completed SLICC/ACR/DI questionnaire at Week 36 visit. 93 subjects received placebo, among them, 83 completed Week 36 visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 82 | 83
scores on a scale | -0.09 (0.59) | -0.17 (0.49)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.3258, student - pooled

8. Secondary Outcome: CLASI Total Activity Change From Baseline at Week 36
Description: Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) was specifically developed to assess the cutaneous manifestations of SLE. It measures both disease activity and permanent damage (e.g. dyspigmentation and scarring) over the entire body surface. CLASI total activity score ranges from 0 to 70, with higher scores indicating more severe skin disease.
Time Frame: Baseline and Week 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 85 | 84
scores on a scale | -3.22 (5.94) | -2.85 (3.60)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.6169, Student - Satterthwaite

9. Secondary Outcome: Number of Participants Who Achieved a Composite SRI-4 Including CS ≤7,5mg/Day at Week 36
Description: SRI (4) plus CS ≤ 7.5 mg/day responder was defined as a participant who had the following criteria at week 36:
  * reduction ≥4 points in SELENA-SLEDAI at week 36 compared with baseline, and
  * no new BILAG A at week 36, and
  * no more than 1 new BILAG B at week 36, and
  * no deterioration in PGA (<10% worsening) on 100-mm VAS compared with baseline plus CS ≤7.5mg equivalent prednisolone per day at week 36
Time Frame: At Week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 79 had CS ≤7,5mg/day at Week 36 visit. 93 subjects received placebo, among them, 77 had CS ≤7,5mg/day at Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 79 | 77
Participants | 46 | 33
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0796, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.932 to 3.524]

10. Secondary Outcome: Number of Participants Who Achieved a Composite SRI-4 Including CS ≤5mg/Day at Week 36
Description: SRI-4 plus CS ≤ 5mg/day responder was defined as a participant who had the following criteria at Week 36:
  * reduction ≥4 points in SELENA-SLEDAI at week 36 compared with baseline, and
  * no new BILAG A at week 36, and
  * no more than 1 new BILAG B at week 36, and
  * no deterioration in PGA (<10% worsening) on 100-mm VAS compared with baseline plus corticosteroids (CS) ≤5mg equivalent prednisolone per day at week 36
Time Frame: At Week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 79 had CS ≤5mg/day at Week 36 visit. 93 subjects received placebo, among them, 77 had CS ≤5mg/day at Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 79 | 77
Participants | 43 | 30
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0762, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.938 to 3.574]

11. Secondary Outcome: Number of Participants With Neutralizing Anti-IFN-alpha Antibodies at W36
Description: Individual serum antibody neutralizing capacity against recombinant IFN-alpha2b was measured by reporter gene assay using Interferon Sensitive Response Element (ISRE) reporter.
Time Frame: At week 36
Population: 91 subjects received IFN-K, among them, 79 were positive for Anti-IFN-alpha antibodies at Week 36 visit.
  No Neutralizing Anti-IFN-alpha antibodies were performed on placebo subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 79 | 0
Participants | 72 | 0

12. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants who reported any treatment-related adverse events until month 9
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 91 | 93
Participants | 75 | 71

13. Other Pre Specified Outcome: CS Mean Daily Dose at W36
Description: mean daily dose of corticosteroid (CS) (prednisone equivalent)
Time Frame: At W36
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 85 | 84
mg/day | 5.42 (3.28) | 7.06 (4.69)
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0097, Student - Satterthwaite

14. Post Hoc Outcome: Number of Participants Who Achieved a Composite SRI-4 (CS ≤5mg/Day) Excluding IFN-K Subjects Without Positive Anti-IFNalpha Neutralizing Antibodies at Week 36
Description: Subjects who had the following criteria defined as : SRI-4 plus CS ≤5mg/day -excluding IFN-K subjects without positive anti-IFN-alpha neutralizing antibodies
Time Frame: At week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 72 had a Composite SRI-4 (CS ≤5mg/day) at Week 36 visit. 93 subjects received placebo, among them, 77 had a Composite SRI-4 CS ≤5mg/day at Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 72 | 77
Participants | 40 | 30
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0425, Pearson's Chi-squared

15. Post Hoc Outcome: Number of Participants Who Achieved a Composite SRI-4 (CS ≤7.5mg/Day) Excluding IFN-K Subjects Without Positive Anti-IFNalpha Neutralizing Antibodies at Week 36
Description: participant who had the following criteria defined as : SRI-4 plus CS ≤7.5mg/day -excluding IFN-K Patients without positive anti-IFN-alpha neutralizing antibodies
Time Frame: At week 36
Population: A total of 185 subjects were randomized and 184 were treated. 91 subjects received IFN-K, among them, 72 had a Composite SRI-4 (CS ≤7.5mg/day) at Week 36 visit. 93 subjects received placebo, among them, 77 had a Composite SRI-4 (CS ≤7.5mg/day) at Week 36 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN-K | Placebo
Number analyzed (Participants) | 72 | 77
Participants | 43 | 33
Statistical Analysis 1: Comparison: IFN-K vs Placebo; Test type: Superiority; p = 0.0396, Pearson's Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) non serious and serious (SAEs) were collected from the start of study Investigational Medicinal Product (IMP) to Week 36.
Description: Due to IFN-K mechanism of action, i.e. immunization, and the administration route, i.e. intramuscular (IM), some AEs, local and/or systemic AEs, were expected and solicited within 7 days after study Investigational Medicinal Product (IMP) administration.
Arm/Group | IFN-K | Placebo
All-Cause Mortality (participants affected / at risk) | 1/91 | 1/93
Serious Adverse Events (participants affected / at risk) | 6/91 | 12/93
Other Adverse Events (participants affected / at risk) | 75/91 | 71/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN-K (N=91) | Placebo (N=93)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Systemic lupus erythematosus (Immune system disorders) | 2 (3) | 3 (3)
Lupus Nephritis (Immune system disorders) | 0 (0) | 1 (1)
Neuropsychiatric Lupus (Immune system disorders) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
chest pain (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Acute respiratory faillure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Postmenauposal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Kaposi's varicelliform eruption (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN-K (N=91) | Placebo (N=93)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 5 (6)
Urinary tract infection (Infections and infestations) | 10 (10) | 9 (10)
Nasopharyngitis (Infections and infestations) | 7 (10) | 2 (2)
Pharyngitis (Infections and infestations) | 6 (7) | 3 (4)
Bronchitis (Infections and infestations) | 5 (5) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 3 (6) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 2 (2)
Cervicitis (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 2 (3) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Vulvovaginitis (Infections and infestations) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (7) | 3 (8)
Pyrexia (General disorders) | 2 (3) | 5 (7)
Injection site pain (General disorders) | 4 (8) | 0 (0)
Injection site induration (General disorders) | 5 (8) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (4)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 2 (2)
Mucosal ulceration (General disorders) | 2 (2) | 1 (1)
Systemic Lupus Erythematosus (Immune system disorders) | 9 (11) | 10 (16)
Systemic Lupus Erythematosus rash (Immune system disorders) | 3 (4) | 3 (4)
Systemic Lupus Erythematosus arthritis (Immune system disorders) | 3 (4) | 4 (4)
Butterfly rash (Immune system disorders) | 1 (2) | 3 (3)
Chronic cutaneous Lupus Erythematosus (Immune system disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (8) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (General disorders) | 2 (2) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Adbominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 10 (19) | 2 (3)
Insomnia (Nervous system disorders) | 3 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Paraesthesia (Nervous system disorders) | 1 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (9) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 4 (5) | 3 (3)
Contusion (Vascular disorders) | 2 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (8)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Conjonctivitis (Eye disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT02665364/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02665364/SAP_001.pdf